CLINICAL TRIAL: NCT06653231
Title: Assessment the Efficacy of Curcumin Local Delivery Gel in Treatment of Periodontitis in Smokers. Randomized Controlled Clinical Trial
Brief Title: Assessment the Efficacy of Curcumin Local Delivery Gel in Treatment of Periodontitis in Smokers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Parryhan Mohamed Abdelsamie, Lecturer of periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102024
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis
Keywords: curcumin; local delivery gel; smokers; periodontitis; RCT
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP with local delivery of Curcumin gel (Experimental): Scaling and root planing in combination with local delivery of Curcumin gel
  Interventions: Drug: local delivery of Curcumin gel
- SRP alone (Active Comparator): Scaling and root plaing alone
  Interventions: Drug: local delivery of Curcumin gel

INTERVENTIONS:
Drug: local delivery of Curcumin gel — The test site will be completely undiluted curcumin gel through a 2 mL disposable syringe was placed in the test site
  Other Names: turmeric plant Curcuma longa L

SUMMARY:
Smokers usually respond less favourably to non-surgical periodontal treatment compared to non-smokers. Numerous studies reported that smoker patients exhibited less reduction in probing depth and less gains in clinical attachment level values following scaling and root planing (Kanmaz et al., 2021, Alwithanani, 2023)

Several studies have proposed the use of adjunctive treatment approaches such as local/systemic antimicrobials and anti-inflammatory agents to improve the effects of basic periodontal therapy in smokers. However, no studies have been published evaluated the conventional management of topically delivered curcumin gel in conjunction with scaling and root planing demonstrating its ability to improve periodontal outcomes in smokers.

Meanwhile, some clinical trials indicate that local and systemic administration of curcumin can enhance the results of SRP in periodontal treatment. Local delivery allows higher concentrations of the active compounds in the diseased site and avoids possible adverse effects of systemic administration.

DETAILED DESCRIPTION:
Tobacco use increases the risk and progression of periodontitis by multiple factors including decreased gingival perfusion, which restricts nutrients and oxygen delivery as well as the removal of waste products. In addition, it affects the circulating levels of immune-inflammatory cells in gingival crevicular fluid, and affects the dysbiosis microbiota reducing the ability of the periodontium to repair.

Curcumin is an extract from the turmeric plant Curcuma longa L. It has been shown potent anti-microbial, anti-carcinogenic, antiviral, antioxidant, and anti-inflammatory properties.

In periodontitis, curcumin plays a pivotal role in anti-inflammatory properties, by inhibiting pro-inflammatory cytokines, reducing the prostaglandin biosynthesis, inhibiting the mRNA and protein expression of cyclo-oxygenase-2, through down-regulation of NF-kB activation.

Meanwhile, some clinical trials indicate that local and systemic administration of curcumin can enhance the results of SRP in periodontal treatment; local delivery allows higher concentrations of the active compounds in the diseased site and avoids possible adverse effects of systemic administration (Pérez-Pacheco et al., 2021, Borgohain et al., 2023, Chatzopoulos et al., 2023).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with generalized periodontitis with stage II
2. Nonsurgical or surgical periodontal therapy in the last 3 months were considered as eligible for the study.
3. Current smoker or smoker over the past 5 years.

Exclusion Criteria:

1. Presence of overhanging restorations,
2. antibiotics or any form of periodontal therapy in the previous 6 months.
3. History of systemic disease, cardiovascular diseases, diabetes mellitus, hypertension, bleeding disorders, hyperparathyroidism, and compromised medical conditions, pregnancy and lactation.
4. Teeth with both endo-perio lesions.
5. Patient on antibiotics within 3 months prior to the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — age group between 21 and 50 years
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | 45 days
  The depth of the pocket will be measured from the gingival margin to the base of the pocket.
clinical attachment level | 45 days
  The clinical attachment level will be measured from the CEJ to the base of pocket.

SECONDARY OUTCOMES:
gingival index | 45 days
  Score 0 normal gingiva and no inflammation Score 1 mild inflammation with a slight change in colour, slight oedema, no bleeding on probing.
  Score 2 moderate inflammation with redness, oedema and glazing or bleeding on probing.
  Score 3 severe inflammation with marked redness and hypertrophy and a tendency toward spontaneous bleeding and ulceration.
Paque index | 45 days
  Score 0 no plaque Score 1 A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which cannot be seen with the naked eye but only by using disclosing solution or probe.
  Score 2 Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen with the naked eye.
  Score 3 Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin

CONTACTS AND LOCATIONS:
Overall Officials: Parryhan M Abdelsamie, Principal Investigator — MTI University
Locations (1):
- MTI University, Cairo, Egypt